CLINICAL TRIAL: NCT06582121
Title: Controlled, Multicenter Study of Sleep Disorders in Prodromal and Definite Parkinsons Disease
Brief Title: Study of Sleep Disorders in Prodromal and Definite Parkinsons Disease
Acronym: SOMPARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230127
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; REM Sleep Behavior Disorder (iRBD)
Keywords: Parkinson disease; isolated RBD; Sleep
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder | interventions — Biological Factors; Urination; Blood Specimen Collection; Defecation

STUDY DESIGN:
Intervention Model Description: All participant will do polysomnographies during a 2-days stay in hospital with electroencephalogram, electromyogram and questionnaries. The urine will be also collected during 2 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): Study of the sleep with polysomnography during a 2-days stay in hospital. Other exam will be done during the 2 days.
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — An overnight sleep study
  Other Names: Biology (urine, blood, faeces); Questionnaries; electromyogram; electroencephalogram

SUMMARY:
Multicenter controlled study of sleep disorders in isolated REM Behavior Disorder and Parkinson's disease (SOMPARK)

DETAILED DESCRIPTION:
Sleep disturbances are common and understudied in established or prodromal Parkinson's disease. The purpose of this study is to systematically and comprehensively determine the clinical characteristics and electrophysiologic patterns of the major sleep disorders in PD and isolated RBD.

ELIGIBILITY:
Inclusion Criteria:

Common to all groups:

* Age superior 18 years
* Patients who have received complete information about the study from an investigator and who fully consent to participate.

For Parkinson Disease (PD):

* Patients followed for PD diagnosed according to international criteria for the diagnosis of PD (MDS criteria),
* A MoCA score greater than 20/30
* No treatment with deep brain stimulation.

For REM Sleep Behavior Disorder (RBD):

* Diagnosis of RBD according to ICSD-3 criteria: presence on polysomnography of an abnormal elevation of muscle tone during REM sleep (more than 18% of REM sleep without chin atonia) and/or the presence of REM sleep behaviors on video-polysomnography,
* Absence of progressive neurodegenerative pathology: absence of diagnostic criteria for PD, multiple system atrophy, or Lewy body dementia.

For healthy controls:

- No neurological or psychiatric disease

Exclusion Criteria:

Common to all groups:

* Pregnant or breastfeeding women
* Subjects under guardianship/conservatorship
* Persons deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 457 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Polysomnography to compare sleep efficiency | 25 months
  Using polysomnography to compare sleep efficiency in the 3 study populations during the first night

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Lille, Lille
  - CHU de Lyon, Lyon
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - CHU Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No